CLINICAL TRIAL: NCT02548715
Title: Levothyroxine Treatment of Subclinical Hypothyroidism After Non-thyroid Head and Neck Surgery: A Randomized Controlled Trial
Brief Title: Levothyroxine Treatment for Subclinical Hypothyroidism After Head and Neck Surgery
Acronym: LSHT
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00043413
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Hypothyroidism; Neoplasms; Postoperative Complications
Keywords: thyroxine; Otolaryngology
MeSH Terms: conditions — Hypothyroidism; Neoplasms; Postoperative Complications | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Daily placebo
  Interventions: Drug: Placebo
- Treatment (Experimental): Participants administered daily levothyroxine at 1.6mcg/kg to a target normal TSH, measured at 6 weeks after the initiation of therapy
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine
  Other Names: Synthroid
  Arms: Treatment
Drug: Placebo
  Arms: Control

SUMMARY:
Patients that require treatment for cancers of the head and neck often require a combination of surgery and/or radiation and chemotherapy. Hypothyroidism is one of the most common complications, and has been associated with post-operative complications such as wound healing problems, fistula formation, and decreased quality of life and survival. Several studies have examined hypothyroidism after radiation to the head and neck, but few have examined this after non-thyroid head and neck surgery. Head and neck resection is theorized to devascularize the thyroid, thus resulting in post-operative hypothyroidism.

Synthroid is a synthetic thyroid hormone often used in cases of patients with proven hypothyroidism and after surgical thyroid removal. It's use has been in effect and studied for over fifty years.

Treatment algorithms for hypothyroidism are well published. However, treatment of subclinical hypothyroidism (elevated TSH with normal or near-normal T3/T4) is controversial. The rate of subclinical hypothyroidism after non-thyroid head and neck surgery is high (up to 20%), and is associated with post-operative complications as noted above.

Therefore the investigators propose a double blinded randomized controlled trial comparing outcomes of patients that develop subclinical hypothyroidism after head and neck surgery, who are given a standardized dose of synthroid treatment versus those treated with placebo. The main outcomes to be examined are post-operative complications (wound healing issues, fistula formation), survival, and quality of life measures.

DETAILED DESCRIPTION:
Background and Scope:

Hypothyroidism is one of the most common complications following multimodality treatment for head and neck cancer, with an incidence of 7-58% depending on the subsite. The causes for this high rate of hypothyroidism following treatment for head and neck cancer are multifactorial. Patients treated for head and neck cancer often require radiation therapy (RT). The negative effects of RT on the thyroid are well published, and the resultant hypothyroidism can have widespread implications on a patient's physical and mental health. Head and neck surgery has also been hypothesized to devascularize and disturb the overall anatomical structure of the thyroid, thus contributing to the high incidence of hypothyroidism after surgery.

Despite the literature demonstrating the connection between head and neck cancer treatment and hypothyroidism, complications from this illness after major head and neck surgery remain common. Decreased survival as well as increased rates of fistulas, infections, and wound breakdown are some of the physical consequences. Other possible issues include decreased functional outcomes and increased mental illness, as these are known consequences of untreated hypothyroidism. While several studies have examined the rate and timing of hypothyroidism after radiation to the head and neck, there is a paucity of literature on the effect of surgery on thyroid function. Specifically, in patients treated with single modality surgery, and in patients treated with primary surgery before the start of RT, when the risk of wound complications is high.

Synthroid is a synthetic thyroid hormone, and is the mainstay of treatment of patients with proven hypothyroidism and after surgical thyroid removal. Its use has been in effect and studied for over fifty years. Side effects of the drug most commonly occur with overdosing and will mimic those of hyperthyroidism, which may include: heart palpitations, abdominal pain, nausea, anxiety, confusion, agitation, insomnia, weight loss, and increased appetite. There is a low chance (< 1%) of allergic reaction to the drug, which may include shortness of breath, swelling of the face and tongue.

Whereas treatment algorithms for clinical hypothyroidism are well established, treatment of subclinical hypothyroidism remains controversial. Subclinical hypothyroidism refers to a state of elevated thyroid stimulating hormone (TSH), with normal or near-normal thyroid hormone levels (T3 and T4), or a lack of symptoms of hypothyroidism. Endocrinologists disagree on whether this disease should be treated, since it is almost always asymptomatic, and the treatment is mainly for relief of symptoms. Head and neck cancer patients, however, represent a special population, in which the effects of subclinical hypothyroidism can result in consequences besides symptoms, such as wound healing issues and fistula development as described above. Studies have shown that the rate of subclinical hypothyroidism during head and neck cancer treatment is high.

Therefore the investigators propose a single blinded randomized controlled trial comparing outcomes of patients with subclinical hypothyroidism, who are given a standardized dose of synthroid treatment after head and neck surgery versus those treated with conventional therapy. A secondary goal of this study is to determine the rate of clinical and subclinical hypothyroidism after surgical treatment for head and neck cancer, without RT or before the start of RT.

Objectives:

Primary Objectives:

* To assess the effect synthroid treatment in patients with subclinical hypothyroidism following head and neck surgery and it's effects on survival, gastrostomy tube (G-tube) rates, fistula formation, wound breakdown, and infection.

Secondary Objectives

* To determine the rate of clinical and subclinical hypothyroidism after surgery for head and neck cancer
* To determine the factors that are predictive of the development of clinical and subclinical hypothyroidism after surgery for head and neck cancer

Methods:

This is a single-center double blinded randomized placebo-controlled trial of the effects of synthroid treatment immediately after surgery for head and neck cancer. Patient meeting eligibility criteria will be identified at the time of booking for surgery and approached by a member of the research team.

Data will be collected from the medical records on the variables under study in study-specific data sheets. Data sheets will then be de-identified and input into a secure database that will be password protected hard drive in a room that is locked. Data will then be exported for statistical analysis when collection is complete.

The population will be comprised of patients who underwent surgery with or without a combination of RT and/or chemotherapy for the treatment of non-thyroid head and neck cancer. Surgery is defined as surgical resection with primary closure or reconstruction with loco-regional flaps or autogenous free tissue transfer. RT is defined as curative dose therapy. Chemotherapy is defined as any single agent therapy or combination of cisplatin or carboplatin. Patients will be prospectively enrolled starting from March 1, 2015 until March 1, 2016. The expected accrual of this patient group will be 200 patients. The demographics of head and neck mucosal cancers indicate that the male : female ratio will be 3 : 1 and the mean age will be approximately 60 years with a range of 18 - 85 years.

In order to assess pre- and post-operative thyroid function, each patient will undergo blood testing including TSH, free T3, and free T4 levels one week prior to surgery, and weekly following surgery, up to 8 weeks post-operatively (if not receiving radiation), or until 8 weeks after the start of radiation (if receiving radiation therapy).

Patients will be classified into "normal" (normal TSH and normal free T3 and free T4 levels), "hypothyroid" (elevated TSH, decreased free T3 and free T4), or "subclinical hypothyroid" (elevated TSH (4-10mIU/L), normal free T3 and free T4).

Patients with "normal" thyroid function will not be randomized to any treatment arm, but their post-operative outcomes will be recorded, according to section 8.0. Patients who are "hypothyroid" will be treated for their hypothyroidism according to the standard of care, in keeping with American Thyroid Association (ATA) / American Association of Clinical Endocrinologists (AACE) guidelines.

Patients with "subclinical hypothyroidism" will be randomized to either the treatment arm or placebo arm, at the time of discovery of subclinical hypothyroidism (lab value abnormalities as noted above). Patients who are randomized to the treatment arm will be treated with a standard dose of 1.6mcg/kg/day of synthroid, and the target of treatment will be a normalized TSH (0.2-4.0mIU/L), measured at 6 weeks after treatment, according to ATA/AACE guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven head and neck cancer, as defined by AJCC staging system
* Treated with surgery in Edmonton, Alberta
* Treated with curative intent
* Diagnosis of sub-clinical hypothyroidism after head and neck surgery (TSH 4-10mIU/L, and free T4 10-24pmol/L)

Exclusion Criteria:

* Head and neck cancer of the thyroid gland, or other subsite involving the thyroid gland
* Underwent previous treatment for a different head and neck cancer
* History of radiation therapy and or chemotherapy to the head and neck
* History of thyroid disease as follows:
* Hypothyroidism
* Hyperthyroidism
* Autoimmune thyroid disease including Grave's disease and Hashimoto's thyroiditis
* History of thyroiditis
* History of diabetes mellitus
* History of long term steroid usage
* History of immunocompromise
* History of thyroid surgery
* History of ischemic heart disease
* Age >80
* Patients taking a medication that may alter the metabolism or interact with levothyroxine, which they cannot safely stop (see Appendix A).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a post-operative wound complication | 12 weeks post-operatively
  * Rate of fistula formation
  * Rate of wound breakdown
  * Rate of post-operative infection
  * Rate of flap failure (dehiscence and/or necrosis requiring salvage)

SECONDARY OUTCOMES:
Number of surviving patients at 6 months | 6 months post-operatively
  Disease-free, disease-specific, and overall survival
Number of patients with G-tube | 12 weeks post-operatively
Quality of life based on EQ-5D7 | 12 weeks post-operatively
Number of patients with clinical depression | 12 weeks post-operatively